CLINICAL TRIAL: NCT00392015
Title: A Two Part Clinical Trial Assessing the Safety, Tolerability, Immunogenicity and Protective Efficacy of NMRC-M3V-Ad-PfCA, a Multivalent, Adenovirus-Vectored Plasmodium Falciparum Malaria Vaccine, in Healthy, Malaria-Naïve Adults
Brief Title: NMRC-M3V-Ad-PfCA Vaccine - Clinical Trial 1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency); Military Infectious Diseases Research Program (MIDRP) (Network); Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: S-15-25; HSRRB A-13453 (Other: WRAIR); NMRC.2006.0001 (Other: NMRC)
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Results first posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-04

CONDITIONS: Plasmodium Falciparum
Keywords: Malaria Vaccine; Adenovirus; Plasmodium falciparum
MeSH Terms: conditions — Malaria, Falciparum; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose-escalation (Experimental): NMRC-M3V-Ad-PfCA
  Interventions: Biological: NMRC-M3V-Ad-PfCA
- Regimen-comparison (Experimental): NMRC-MV-Ad-PfC, NMRC-M3V-Ad-PfCA
  Interventions: Biological: NMRC-MV-Ad-PfC, NMRC-M3V-Ad-PfCA

INTERVENTIONS:
Biological: NMRC-M3V-Ad-PfCA — Malaria Vaccine
  Arms: Dose-escalation
Biological: NMRC-MV-Ad-PfC, NMRC-M3V-Ad-PfCA — Malaria Vaccines
  Arms: Regimen-comparison

SUMMARY:
The purpose of this study is to determine whether a new investigational malaria vaccine is safe, well tolerated and effective against experimental exposure to malaria when given to healthy people with no previous exposure to malaria. The vaccine consists of a modified form of a relatively common virus, adenovirus, that has been rendered incapable of replicating itself and modified to deliver the malaria gene of interest to the body's cells allowing the cell to manufacture the protein encoded by the gene and present it to the body's immune system in a more natural and presumably effective way.

DETAILED DESCRIPTION:
The vaccine, called NMRC-M3V-Ad-PfCA (key: NMRC + Multi-antigen Multi-stage, Malaria Vaccine + Adenovectored + P. falciparum CSP & AMA1 antigens), is a combination of two recombinant adenovirus-derived constructs (adenovectors), one expressing the pre-erythrocytic stage antigen circumsporozoite protein (CSP) and the other expressing the erythrocytic stage antigen Apical Membrane Antigen 1 (AMA1), both from the 3D7 strain of P. falciparum. The vector is an attenuated, replication-deficient adenovirus derived from wildtype serotype 5 adenovirus through the deletion of several genes. The vaccine is formulated in a buffered saline solution (Final Formulation Buffer = FFB).

This is a Phase 1/2a, randomized, open-label, dose-escalating trial of the NMRC-M3V-Ad-PfCA vaccine administered intramuscularly to healthy, malaria-naïve adult volunteers. All volunteers will be seronegative (< 1:500, by a luciferase-based neutralizing antibody assay; VRC, Bethesda) for adenovirus serotype 5. In the first part of the study (dose-escalation phase, Part A), 1 x 10^10 particle units (pu) per construct or 2 x 10^10 pu total will be administered to six volunteers as a single dose to assess safety, and 4 weeks later, 5 x 10^10 pu per construct or 1 x 10^11 pu total dose (five-fold dose escalation) will be administered to six additional volunteers. In the second part of the study (regimen-comparison phase, Part B), three regimens for administration will be compared: one dose, two doses administered ten days apart, and two doses administered 16 weeks apart. Separate groups will receive one dose of the individual components of the vaccine (NMRC-MV-Ad-PfC and NMRC-MV-Ad-PfA). Following immunization, volunteers participating in the regimen-comparison phase as well as several non-immunized control volunteers (serving as infectivity controls) will be challenged with P. falciparum sporozoites in order to assess vaccine efficacy against non-immunized controls challenged at the same time. The proposed design of the regimen-comparison phase will provide information to direct selection of an appropriate dosing regimen for subsequent studies, and will also indicate whether the two constituent antigens, when co-formulated, act synergistically, independently, or interfere with each other in the induction of antigen-specific immune responses and protective immunity.

ELIGIBILITY:
INCLUSION CRITERIA:

* Between the ages of 18-50 (inclusive)
* Negative results of HIV ELISA, HbSAg, anti-HCV antibody, and no other clinically significant abnormal laboratory results from screening.
* Adenovirus serotype 5 (Ad5) titer <1:500
* Able to provide written informed consent.
* Complete an Assessment of Understanding and verbalize an understanding of any questions answered incorrectly.
* In good general health without clinically significant medical history or physical exam abnormalities at screening.
* Willing to continue immunogenicity and clinical follow-ups for one year and telephone or mail (electronic/U.S. Postal) contact as long term safety monitoring provision for an additional four years (totaling five years of participation; immunized volunteers only).
* Male and female participants being immunized and female participants being challenged agree to use effective means of birth control (an FDA approved contraceptive, abstinence) between screening and 60 days following last clinical study visit or able to provide evidence of no reproductive capability.

EXCLUSION CRITERIA:

* Have a history of malaria infection, exposure to malaria infection(i.e. you have been to an area that has malaria within the past two years),lived in a country with malaria for more than 5 years or receipt of certain candidate malaria vaccines
* Known immune system disease
* Known blood, heart, liver, kidney disease
* At known significant risk for developing heart disease
* A positive result on HIV testing at screening
* A positive result on Hepatitis B or C testing at screening
* Removal of your spleen
* Taking medication that suppresses the immune system within 30 days of immunization.
* Received or will be receiving another vaccine within 30 days of immunization
* Received blood products (e.g. transfused with blood cells, platelets, plasma or serum) within 120 days of the immunization
* Have had serious adverse reactions to other vaccines including hives, anaphylaxis, respiratory difficulty, tongue/mouth/neck/throat/body swelling or abdominal pain
* Pregnant, breastfeeding, or planning to become pregnant during the next year
* Plan to participate (or have participated in the last 30 days) in any other research study including an investigational drug or device
* Unwilling or unable to participate/complete all study elements
* Evidence of previous infection with adenovirus 5 or prior receipt of an adenovirus containing vaccine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2006-10-12 (Actual); Primary Completion 2016-06-02 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Tamminga, MD, MPH, Principal Investigator — Naval Medical Research Center
Locations (1):
- Naval Medical Research Center (NMRC) Clinical Trials Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ophorst OJ, Radosevic K, Havenga MJ, Pau MG, Holterman L, Berkhout B, Goudsmit J, Tsuji M. Immunogenicity and protection of a recombinant human adenovirus serotype 35-based malaria vaccine against Plasmodium yoelii in mice. Infect Immun. 2006 Jan;74(1):313-20. doi: 10.1128/IAI.74.1.313-320.2006. PMID 16368986
- [Background] Li S, Locke E, Bruder J, Clarke D, Doolan DL, Havenga MJ, Hill AV, Liljestrom P, Monath TP, Naim HY, Ockenhouse C, Tang DC, Van Kampen KR, Viret JF, Zavala F, Dubovsky F. Viral vectors for malaria vaccine development. Vaccine. 2007 Mar 30;25(14):2567-74. doi: 10.1016/j.vaccine.2006.07.035. Epub 2006 Aug 1. PMID 16914237
- [Background] Rodrigues EG, Zavala F, Nussenzweig RS, Wilson JM, Tsuji M. Efficient induction of protective anti-malaria immunity by recombinant adenovirus. Vaccine. 1998 Nov;16(19):1812-7. doi: 10.1016/s0264-410x(98)00181-9. PMID 9795385
- [Derived] Sedegah M, Peters B, Hollingdale MR, Ganeshan HD, Huang J, Farooq F, Belmonte MN, Belmonte AD, Limbach KJ, Diggs C, Soisson L, Chuang I, Villasante ED. Vaccine Strain-Specificity of Protective HLA-Restricted Class 1 P. falciparum Epitopes. PLoS One. 2016 Oct 3;11(10):e0163026. doi: 10.1371/journal.pone.0163026. eCollection 2016. PMID 27695088
- [Derived] Aguiar JC, Bolton J, Wanga J, Sacci JB, Iriko H, Mazeika JK, Han ET, Limbach K, Patterson NB, Sedegah M, Cruz AM, Tsuboi T, Hoffman SL, Carucci D, Hollingdale MR, Villasante ED, Richie TL. Discovery of Novel Plasmodium falciparum Pre-Erythrocytic Antigens for Vaccine Development. PLoS One. 2015 Aug 20;10(8):e0136109. doi: 10.1371/journal.pone.0136109. eCollection 2015. PMID 26292257
- [Derived] Sedegah M, Hollingdale MR, Farooq F, Ganeshan H, Belmonte M, Huang J, Abot E, Limbach K, Chuang I, Tamminga C, Epstein JE, Villasante E. Controlled Human Malaria Infection (CHMI) differentially affects cell-mediated and antibody responses to CSP and AMA1 induced by adenovirus vaccines with and without DNA-priming. Hum Vaccin Immunother. 2015;11(11):2705-15. doi: 10.1080/21645515.2015.1019186. Epub 2015 Aug 20. PMID 26292027
- [Derived] Sedegah M, Hollingdale MR, Farooq F, Ganeshan H, Belmonte M, Kim Y, Peters B, Sette A, Huang J, McGrath S, Abot E, Limbach K, Shi M, Soisson L, Diggs C, Chuang I, Tamminga C, Epstein JE, Villasante E, Richie TL. Sterile immunity to malaria after DNA prime/adenovirus boost immunization is associated with effector memory CD8+T cells targeting AMA1 class I epitopes. PLoS One. 2014 Sep 11;9(9):e106241. doi: 10.1371/journal.pone.0106241. eCollection 2014. PMID 25211344
- [Derived] Tamminga C, Sedegah M, Maiolatesi S, Fedders C, Reyes S, Reyes A, Vasquez C, Alcorta Y, Chuang I, Spring M, Kavanaugh M, Ganeshan H, Huang J, Belmonte M, Abot E, Belmonte A, Banania J, Farooq F, Murphy J, Komisar J, Richie NO, Bennett J, Limbach K, Patterson NB, Bruder JT, Shi M, Miller E, Dutta S, Diggs C, Soisson LA, Hollingdale MR, Epstein JE, Richie TL. Human adenovirus 5-vectored Plasmodium falciparum NMRC-M3V-Ad-PfCA vaccine encoding CSP and AMA1 is safe, well-tolerated and immunogenic but does not protect against controlled human malaria infection. Hum Vaccin Immunother. 2013 Oct;9(10):2165-77. doi: 10.4161/hv.24941. Epub 2013 Jun 4. PMID 23899517
- [Derived] Tamminga C, Sedegah M, Regis D, Chuang I, Epstein JE, Spring M, Mendoza-Silveiras J, McGrath S, Maiolatesi S, Reyes S, Steinbeiss V, Fedders C, Smith K, House B, Ganeshan H, Lejano J, Abot E, Banania GJ, Sayo R, Farooq F, Belmonte M, Murphy J, Komisar J, Williams J, Shi M, Brambilla D, Manohar N, Richie NO, Wood C, Limbach K, Patterson NB, Bruder JT, Doolan DL, King CR, Diggs C, Soisson L, Carucci D, Levine G, Dutta S, Hollingdale MR, Ockenhouse CF, Richie TL. Adenovirus-5-vectored P. falciparum vaccine expressing CSP and AMA1. Part B: safety, immunogenicity and protective efficacy of the CSP component. PLoS One. 2011;6(10):e25868. doi: 10.1371/journal.pone.0025868. Epub 2011 Oct 7. PMID 22003411
- [Derived] Sedegah M, Tamminga C, McGrath S, House B, Ganeshan H, Lejano J, Abot E, Banania GJ, Sayo R, Farooq F, Belmonte M, Manohar N, Richie NO, Wood C, Long CA, Regis D, Williams FT, Shi M, Chuang I, Spring M, Epstein JE, Mendoza-Silveiras J, Limbach K, Patterson NB, Bruder JT, Doolan DL, King CR, Soisson L, Diggs C, Carucci D, Dutta S, Hollingdale MR, Ockenhouse CF, Richie TL. Adenovirus 5-vectored P. falciparum vaccine expressing CSP and AMA1. Part A: safety and immunogenicity in seronegative adults. PLoS One. 2011;6(10):e24586. doi: 10.1371/journal.pone.0024586. Epub 2011 Oct 7. PMID 22003383

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: NMRC-M3V-Ad-PfCA, 2x10^10 pu; Group 2: NMRC-M3V-Ad-PfCA, 1x10^11 pu: Part A is a dose escalation of NMRC-M3V-Ad-PfCA (2 antigen combination) using 2 dose groups: Group 1 received a single low dose of 2x10^10 pu and Group 2 received a single high dose of 1x10^11 pu. Injections were staggered by 4 weeks in order to assess the safety and tolerability of the vaccine and define the dose to be used in Part B.
- Group 3: NMRC-M3V-Ad-PfCA, 2x10^10 pu; Group 4: NMRC-MV-Ad-PfC, 1x10^10 pu: Part B is the challenge phase to assess protective efficacy. Subjects in part B received 2 intramuscular injections given 16 weeks apart: Group 3 NMRC-M3V-Ad-PfCA (2 antigen combination) at a dose of 2x10^10 pu, or Group 4 NMRC-MV-Ad-PfC (single antigen) at 1x10^10 pu dose. Infectivity control subjects were challenged with Group 3 and Group 4.
- Group 3: Infectivity Control: Infectivity control subjects were challenged with Group 3
- Group 4: Infectivity Control: Infectivity control subjects were challenged with Group 4
Period: Overall Study
Arm/Group | Group 1: NMRC-M3V-Ad-PfCA, 2x10^10 pu | Group 2: NMRC-M3V-Ad-PfCA, 1x10^11 pu | Group 3: NMRC-M3V-Ad-PfCA, 2x10^10 pu | Group 3: Infectivity Control | Group 4: NMRC-MV-Ad-PfC, 1x10^10 pu | Group 4: Infectivity Control
Started | 6 | 6 | 20 | 6 | 15 | 6
Completed | 4 | 6 | 16 | 5 | 12 | 6
Not Completed | 2 | 0 | 4 | 1 | 3 | 0
Not completed — Lost to Follow-up | 2 | 0 | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Previous trial recipient | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 2: NMRC-M3V-Ad-PfCA,1x10^11 pu: Part A is a dose escalation of NMRC-M3V-Ad-PfCA (2 antigen combination) using 2 dose groups: Group 1 received a single low dose of 2x10^10 pu and Group 2 received a single high dose of 1x10^11 pu. Injections were staggered by 4 weeks in order to assess the safety and tolerability of the vaccine and define the dose to be used in Part B.
- Group 3: Infectivity Control; Group 4: Infectivity Control: Infectivity control subjects were challenged with Group 3 and Group 4
- Total: Total of all reporting groups
Arm/Group | Group 1: NMRC-M3V-Ad-PfCA, 2x10^10 pu | Group 2: NMRC-M3V-Ad-PfCA,1x10^11 pu | Group 3: NMRC-M3V-Ad-PfCA, 2x10^10 pu | Group 3: Infectivity Control | Group 4: NMRC-MV-Ad-PfC, 1x10^10 pu | Group 4: Infectivity Control | Total
Number analyzed (Participants) | 6 | 6 | 20 | 6 | 15 | 6 | 59
Age, Customized [Count of Participants; unit: Participants]
  18-20 years | 0 | 1 | 2 | 0 | 0 | 0 | 3
  21-30 years | 3 | 2 | 10 | 2 | 4 | 2 | 23
  31-40 years | 2 | 1 | 3 | 3 | 6 | 1 | 16
  41-50 years | 1 | 2 | 5 | 1 | 5 | 3 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 6 | 2 | 4 | 3 | 20
  Male | 5 | 2 | 14 | 4 | 11 | 3 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 1 | 1 | 0 | 6
  Not Hispanic or Latino | 5 | 6 | 17 | 5 | 14 | 6 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Asian/Pacific Islander fall under one category in the study and the number of participants in this category are noted under Asian in the baseline measure table
  Participants
    American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Asian | 0 | 0 | 0 | 0 | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 2 | 3 | 9 | 3 | 8 | 1 | 26
    White | 3 | 3 | 7 | 2 | 4 | 5 | 24
    More than one race | 1 | 0 | 3 | 1 | 1 | 0 | 6
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 20 | 6 | 15 | 6 | 59

OUTCOME MEASURES:

1. Primary Outcome: Part A Dose-Escalation: Number of Participants Who Experienced Any Serious Adverse Events Related To Vaccine Administration
Description: To assess the safety and tolerability of NMRC-M3V-Ad-PfCA, in a dose-escalation design (Part A), in healthy malaria-naïve adults. Part A was a dose escalation of NMRC-M3V-AdPfCA (2 antigen combination) using two dose groups, 2x10^10 pu (Group 1) and 1x10^11 pu (Group 2). Subjects received a single intramuscular injection with the injections in the 2 groups staggered by 4 weeks in order to assess the safety and tolerability of the vaccine and define the dose to be used in Part B. The vaccine was to be considered safe and well-tolerated if there were no severe or serious adverse events related to vaccine administration.
Time Frame: Through Study Completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Group 1 received NMRC-M3V-Ad-PfCA (2 antigen combination) at a single low dose of 2x10^10 pu on Week 0
- Group 2: Group 2 received NMRC-M3V-Ad-PfCA (2 antigen combination) at a single high dose of 1x10^11 pu on Week 4.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

2. Primary Outcome: Part B Regimen-Comparison: Number of Participants With Any Serious Adverse Events Related to Vaccine Administration
Description: To assess the safety and tolerability of NMRC-M3V-Ad-PfCA, in a regimen-comparison design (Part B), in healthy malaria-naïve adults. Subjects in part B received 2 intramuscular injections given 16 weeks apart: Group 3 NMRC-M3V-Ad-PfCA (2 antigen combination) at a dose of 2x10^10 pu, or Group 4 NMRC-MV-Ad-PfC (single antigen) at 1x10^10 pu dose. The vaccine was to be considered safe and well-tolerated if there were no severe or serious adverse events related to vaccine administration.
Time Frame: Through Study Completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Group 3: 2 doses of NMRC-M3V-Ad-PfCA (2x10^10 pu) administered intramuscular 16 weeks apart on Week 16 and Week 32
- Group 4: 2 doses of NMRC-MV-Ad-PfC (1x10^10 pu) administered intramuscular 16 weeks apart on Week 16 and Week 32
Arm/Group | Group 3 | Group 4
Number analyzed (Participants) | 20 | 15
Participants | 0 | 0

3. Primary Outcome: Part B Regimen Comparison: Time to Parasitemia to Assess the Protective Efficacy Against Sporozoite Challenge (Pf, 3D7 Strain)
Description: Protective efficacy was assessed by conducting a homologous 3D7 strain sporozoite challenge 3 weeks after the second NMRCMV-Ad-PfC immunization. Time to parasitemia was measured in both vaccinated and unvaccinated volunteers (infectivity controls) in Group 3 (NMRC-M3V-Ad-PfCA (2 antigen combination) at a dose of 2x10^10 pu) and Group 4 (NMRC-MV-Ad-PfC (single antigen) at 1x10^10 pu dose). Infectivity control subjects were challenged with Group 3 and Group 4. Each volunteer was monitored for the onset of signs and symptoms of malaria and by daily Giemsa-stained thick blood films with positive films confirmed by a second reader. The identity of immunized and non-immunized volunteers was known to the clinical trial staff but not to the microscopists reading the malaria smears.
Time Frame: Through Study Completion, an average of 1 year
Measure: Geometric Mean (Full Range); unit: days
Groups:
- Group 3: 2 doses of NMRC-M3V-Ad-PfCA (2x10^10 pu) administered intramuscular 16 weeks apart on Week 16 and Week 32 followed by a sporozoite challenge 3 weeks later. Infectivity control subjects (not vaccinated) were also challenged.
- Group 3 Infectivity Control; Group 4 Infectivity Control: Infectivity control subjects (not vaccinated) were also challenged
- Group 4: 2 doses of NMRC-MV-Ad-PfC (1x10^10 pu) administered intramuscular 16 weeks apart on Week 16 and Week 32 followed by a sporozoite challenge 3 weeks later. Infectivity control subjects (not vaccinated) were also challenged.
Arm/Group | Group 3 | Group 3 Infectivity Control | Group 4 | Group 4 Infectivity Control
Number analyzed (Participants) | 20 | 6 | 15 | 6
days | 12.1 [9 to 16] | 11.8 [11 to 13] | 13.37 [12 to 16] | 12.96 [12 to 14]

4. Secondary Outcome: Part A Dose-Escalation: To Assess the Immunogenicity of NMRC-M3V-Ad-PfCA in Healthy Malaria-Naïve Adults Using ELISpot IFN-γ Responses
Description: The NMRC-M3V-Ad-PfCA vaccine combines two adenovectors encoding circumsporozoite protein (CSP) and apical membrane antigen-1 (AMA1). In Group 1 healthy volunteers received one intramuscular injection of 2x10^10 pu at Week 0 and in Group 2 a five-fold higher dose of 1 x 10^11 pu at Week 4. Immunogenicity was assessed by ELISpot IFN-γ responses against synthetic peptides derived from CSP and AMA1 as the range of spot forming cells/million peripheral blood mononuclear cells [sfc/m].
Time Frame: One month post immunization
Measure: Geometric Mean (Full Range); unit: sfc/m
Groups:
- Circumsporozoite Protein (CSP); Apical Membrane Antigen-1 (AMA1): The NMRC-M3V-Ad-PfCA vaccine combines two adenovectors encoding circumsporozoite protein (CSP) and apical membrane antigen-1 (AMA1)
Arm/Group | Circumsporozoite Protein (CSP) | Apical Membrane Antigen-1 (AMA1)
Number analyzed (Participants) | 6 | 6
sfc/m
  Group 1 | 422 [422 to 337] | 862 [862 to 697]
  Group 2 | 154 [154 to 203] | 423 [423 to 466]

5. Secondary Outcome: Part B Regimen-Comparison: To Assess the Immunogenicity of NMRC-M3V-Ad-PfCA in Healthy Malaria-Naïve Adults Using ELISpot IFN-γ Responses in Group 3
Description: The NMRC-M3V-Ad-PfCA vaccine combines two adenovectors encoding circumsporozoite protein (CSP) and apical membrane antigen-1 (AMA1). Group 3 healthy volunteers received 2 intramuscular injections of NMRC-M3V-Ad-PfCA (2 antigen combination) at a dose of 2x10^10 pu at Week 16 and Week 32. Immunogenicity was assessed by ELISpot IFN-γ responses against synthetic peptides derived from CSP and AMA1 using peripheral blood mononuclear cells during the study. IFN-γ ELISpot responses were measured as the range of spot forming cells/million peripheral blood mononuclear cells [sfc/m].
Time Frame: 22-23 days post immunization
Measure: Geometric Mean (Full Range); unit: sfc/m
Arm/Group | Circumsporozoite Protein (CSP) | Apical Membrane Antigen-1 (AMA1)
Number analyzed (Participants) | 20 | 20
sfc/m | 273 [38 to 2550] | 1303 [435 to 4594]

6. Secondary Outcome: Part B Regimen-Comparison: To Assess the Immunogenicity of NMRC-MV-Ad-PfC in Healthy Malaria-Naïve Adults Using ELISpot IFN-γ Responses in Group 4
Description: Group 4 healthy volunteers received 2 intramuscular injections of NMRC-MV-Ad-PfC (single antigen) at a dose of 1x10^10 pu at Week 16 and Week 32. Immunogenicity was assessed by ELISpot IFN-γ responses against synthetic peptides derived from circumsporozoite protein (CSP) using peripheral blood mononuclear cells during the study. IFN-γ ELISpot responses measured as the range of spot forming cells/million peripheral blood mononuclear cells [sfc/m].
Time Frame: 4 weeks post immunization
Measure: Geometric Mean (Full Range); unit: sfc/m
Groups:
- Circumsporozoite Protein (CSP): Synthetic peptides derived from CSP
Arm/Group | Circumsporozoite Protein (CSP)
Number analyzed (Participants) | 15
sfc/m | 323 [71 to 1127]

7. Secondary Outcome: Part A Dose-Escalation: To Assess the Immunogenicity of NMRC-M3V-Ad-PfCA in Healthy Malaria-Naïve Adults Using Intracellular Cytokine Staining of CD4+ and CD8+ T Cell IFN-γ Responses
Description: The NMRC-M3V-Ad-PfCA vaccine combines two adenovectors encoding circumsporozoite protein (CSP) and apical membrane antigen-1 (AMA1). In Group 1 healthy volunteers received one intramuscular injection of 2x10^10 pu at Week 0 and in Group 2 a five-fold higher dose of 1 x 10^11 pu at Week 4. Immunogenicity was assessed by Intracellular Cytokine Staining of CD4+ and CD8+ T cell IFN-γ responses to AMA1 and CSP using peripheral blood mononuclear cells during the study. CD4+ and CD8+ T cell IFN-γ responses were measured as percentage (%) range of positive responses.
Time Frame: One month post immunization
Measure: Geometric Mean (Full Range); unit: percentage of cells
Arm/Group | Circumsporozoite Protein (CSP) | Apical Membrane Antigen-1 (AMA1)
Number analyzed (Participants) | 6 | 6
percentage of cells
  Group 1 (% CD8+) | 0.210 [0.210 to 0.14] | 0.44 [0.44 to 0.58]
  Group 1 (% CD4+) | 0.044 [0.044 to 0.075] | 0.086 [0.086 to 0.17]
  Group 2 (% CD8+) | 0.020 [0.020 to 0.12] | 0.15 [0.15 to 0.46]
  Group 2 (% CD4+) | 0.006 [0.006 to 0.017] | 0.035 [0.035 to 0.038]

8. Secondary Outcome: Part B Regimen-Comparison: To Assess the Immunogenicity of NMRC-M3V-Ad-PfCA in Healthy Malaria-Naïve Adults Using Intracellular Cytokine Staining CD4+ and CD8+ T Cell IFN-γ Responses in Group 3
Description: The NMRC-M3V-Ad-PfCA vaccine combines two adenovectors encoding circumsporozoite protein (CSP) and apical membrane antigen-1 (AMA1). Group 3 healthy volunteers received 2 intramuscular injections of NMRC-M3V-Ad-PfCA (2 antigen combination) at a dose of 2x10^10 pu at Week 16 and Week 32. Immunogenicity was assessed by Intracellular Cytokine Staining of CD4+ and CD8+ T cell IFN-γ responses to AMA1 and CSP measured using peripheral blood mononuclear cells during the study. CD4+ and CD8+ T cell IFN-γ responses were measured as percentage (%) range of positive responses.
Time Frame: 22-23 days post immunization
Measure: Geometric Mean (Full Range); unit: percentage of cells
Arm/Group | Circumsporozoite Protein (CSP) | Apical Membrane Antigen-1 (AMA1)
Number analyzed (Participants) | 20 | 20
percentage of cells
  % CD4+ Cells | 0.030 [0.02 to 0.18] | 0.090 [0.027 to 0.478]
  % CD8+ Cells | 0.093 [0.03 to 0.47] | 0.216 [0.04 to 2.08]

9. Secondary Outcome: Part B Regimen-Comparison: To Assess the Immunogenicity of NMRC-MV-Ad-PfC in Healthy Malaria-Naïve Adults Using Intracellular Cytokine Staining of CD4+ and CD8+ T Cell IFN-γ Responses in Group 4
Description: Group 4 healthy volunteers received 2 intramuscular injections of NMRC-MV-Ad-PfC (single antigen) at a dose of 1x10^10 pu at Week 16 and Week 32. Immunogenicity was assessed by Intracellular Cytokine Staining of CD4+ and CD8+ T cell IFN-γ responses to synthetic peptides derived from circumsporozoite protein (CSP) using peripheral blood mononuclear cells during the study. CD4+ and CD8+ T cell IFN-γ responses were measured as percentage (%) range of positive responses.
Time Frame: 4 weeks post immunization
Measure: Geometric Mean (Full Range); unit: percentage of cells
Arm/Group | Circumsporozoite Protein (CSP)
Number analyzed (Participants) | 15
percentage of cells
  % CD4+ Cells | 0.039 [0.00141 to 0.137]
  % CD8+ Cells | 0.09 [0.012 to 0.556]

ADVERSE EVENTS:
Time Frame: Through Study Completion, an average of 1 year
Description: Occurrence of solicited adverse events over a 14-day follow-up period (day of vaccination and 13 subsequent days) and unsolicited adverse events over a 30 day follow-up period (day of immunization and 29 subsequent days) in vaccinated subjects Groups 1-4. Other (Not Including Serious) Adverse Events were not collected for the infected control group. Serious adverse events during the one year active study period in vaccinated subjects Groups 1-4 and non-vaccinated infectivity control subjects.
Groups:
- Group 1: Single low dose (2x10^10 pu) of NMRC-M3V-Ad-PfCA administered intramuscular on Week 0
- Group 2: Single high dose (1x10^11 pu) of NMRC-M3V-Ad-PfCA administered intramuscular on Week 4
- Group 3: 2 doses of NMRC-M3V-Ad-PfCA (2x10^10 pu) administered intramuscular 16 weeks apart on Week 16 and Week 32 followed by a sporozoite challenge 2 to 4 weeks after the second immunization.
- Group 3 Infectivity Control; Group 4 Infectivity Control: Infectivity Control (not vaccinated) were also challenged
- Group 4: 2 doses of NMRC-MV-Ad-PfC (1x10^10 pu) administered intramuscular 16 weeks apart on Week 16 and Week 32 followed by a sporozoite challenge 2 to 4 weeks after the second immunization.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 3 Infectivity Control | Group 4 | Group 4 Infectivity Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/20 | 1/6 | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/20 | 1/6 | 0/15 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 5/6 | 9/20 | 0/0 | 13/15 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=6) | Group 2 (N=6) | Group 3 (N=20) | Group 3 Infectivity Control (N=6) | Group 4 (N=15) | Group 4 Infectivity Control (N=6)
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Suicide (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=6) | Group 2 (N=6) | Group 3 (N=20) | Group 3 Infectivity Control (N=0) | Group 4 (N=15) | Group 4 Infectivity Control (N=0)
Pain/tenderness (General disorders) | 5 | 5 | 9 | NA | 13 | NA
Erythema (General disorders) | 0 | 0 | 1 | NA | 0 | NA
Induration/swelling (General disorders) | 0 | 1 | 1 | NA | 0 | NA
Warmth (General disorders) | 0 | 1 | 2 | NA | 0 | NA
Hives (General disorders) | 0 | 0 | 1 | NA | 0 | NA
Lymphadenopathy (General disorders) | 2 | 0 | 0 | NA | 0 | NA
Limited arm motion (General disorders) | 1 | 0 | 0 | NA | 0 | NA
Headache (Nervous system disorders) | 2 | 3 | 3 | NA | 2 | NA
Malaise (General disorders) | 1 | 4 | 3 | NA | 2 | NA
Fever (General disorders) | 1 | 4 | 2 | NA | 1 | NA
Chills (General disorders) | 0 | 4 | 2 | NA | 1 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | NA | 2 | NA
Fatigue (General disorders) | 0 | 0 | 5 | NA | 2 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | NA | 0 | NA
Nausea/vomiting (Gastrointestinal disorders) | 2 | 3 | 2 | NA | 2 | NA
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | NA | 2 | NA
Blurred vision (Eye disorders) | 0 | 1 | 0 | NA | 0 | NA
Dizziness (Nervous system disorders) | 0 | 1 | 1 | NA | 1 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | 0 | NA
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | 1 | NA
Pink eye/conjunctivitis D (Eye disorders) | 0 | 0 | 0 | NA | 1 | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | 1 | NA
Eye pain/irritation (Eye disorders) | 0 | 0 | 0 | NA | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No